CLINICAL TRIAL: NCT06076915
Title: Usability and Feasibility Trial of an Exergame-based Occupational Health Intervention at Two Swiss Workforce Companies
Brief Title: Usability and Feasibility of an Occupational Exergame-based Intervention
Acronym: Senso@Work
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Principal Investigator, Eling DeBruin, Prof., Swiss Federal Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: EK-2021-N-49
Record Dates: First submitted 2022-11-15; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Healthy
Keywords: occupational health; cognitive-motor intervention; exergame; well-being

STUDY DESIGN:
Intervention Model Description: The study is designed as a two-arm crossover pilot trial. The 12-week lasting study includes three assessment points (T0, T1, T2). After signing informed consent, participants will be randomly allocated to either group 1 (G1) or group 2 (G2), using simple (unrestricted) randomization based on a random-number table. All participants perform baseline assessments at T0. Depending on their random allocation to group 1 (G1) or group 2 (G2), they will either continue with their usual daily work life (G2), or they will start the intervention period (G1) , where they will implement the exergame training plan in their working schedule. After six weeks, both groups will perform the T1 assessments, and the program will be switched, meaning G2 will perform the exergame training and G1 will have their control period. After completing the intervention at week 12, both groups will perform the final assessments (T2).
Who Masked: Outcomes Assessor
Masking Description: The outcome evaluator of the pre- and post-measurement was blinded to group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G1 (Group 1) (Experimental): Experimental: Exergame Training, then Usual Daily Work
  Participants of G1 first received the Exergame Training (integrated into their working schedule). After 6 weeks, they no longer received exergame training but followed their normal work schedule for another 6 weeks.
  Interventions: Behavioral: Exergame training
- G2 (Group 2) (Experimental): Experimental: Usual Training Work, then Exergame Training
  Participants of G2 first followed their normal work schedule for 6 weeks and then received the Exergame training for another 6 weeks.
  Interventions: Behavioral: Exergame training

INTERVENTIONS:
Behavioral: Exergame training — During the exergame intervention period, the participants in the respective group will be asked to train at least two times per week for 10 minutes per session. The proposed 10 to 15 min-sessions can also be split up into multiple short training slots during the day, to thus reach the targeted 10 minutes. Moreover, the participants are allowed to train even more during their "exergame-intervention" period of six weeks. However, during the control period of six weeks, they are prohibited from training on the device.
  The training program will start with four pre-defined programs of the Dividat Senso (Dividat AG, Schindellegi, Switzerland; CE certification) program. This training program will be adapted weekly by the investigator to generate new stimuli through varying games and thereby also further support the motivation.

SUMMARY:
High levels of sustained sedentary time in office workers are associated with non-communicable diseases as e.g. cardio-vascular diseases or diabetes. Moreover, recent evidence has further suggested a relationship between prolonged sitting periods and adverse mental health outcomes. Based on these facts, various types of occupational health-related interventions have already been undertaken, thereby mostly focusing on physical aspects. However, a promising intervention option that has only rarely been investigated in this context, are so-called exergames, which allow a combined physical and cognitive training in a motivating and time-efficient manner. This pilot trial aims to determine the usability and feasibility of an exergame-based intervention targeting occupational health aspects, whilst secondarily exploring potential effects on physical and cognitive functions.

The study is planned for healthy (self-reported) office workers, aged between 18 and 65 years. Participants are asked to perform a minimum of 18 training sessions with a duration of 10-20 minutes during a period of six weeks. The design is planned as a two-arm crossover trial, where participants will randomly get allocated to a group, and either start with the training period or the control period (no training). After having completed the six-week training period, participants will evaluate the usability and report their experience with the exergame device. In terms of evaluation of the feasibility, adherence and attrition rates will be calculated at the end of the study. Before, after six weeks, as well as after 12 weeks, cognitive and physical assessments will be performed and questionnaires on behalf of stress experience and management will be elicited.

The findings of this pilot trial will help to explore the possibilities of designing occupational health interventions by the implementation of motor-cognitive exergames. In addition, this trial offers the possibility of exploratorily analyzing the effects of exergame training in office-workers.

DETAILED DESCRIPTION:
Office workers spend around 65-75% of their working hours in a seated position, whereby more than 50% of this time is accumulated in prolonged periods of sustained sitting. Growing evidence has shown, that such prolonged periods of sitting have deleterious health effects, even in adults meeting the usual physical activity guidelines of 150 minutes of weekly physical activity. These negative health effects include cardiovascular disease, general higher all-cause mortality and diabetes, whose strength of association is the most consistent. Moreover, sedentary behavior is negatively associated with reduced cognitive functions, whereby the associations are largely dependent on the assessed outcomes. Reducing sedentary phases by implementing intermittent physical activity was reported providing beneficial effects on multiple systems that are relevant for brain health, such as blood pressure, sympathetic function, or vascular function.

In addition to these direct physical consequences of working seated in an office, occupational stress can exert a further negative influence on employees. Such persisting increased levels of stress can lead to high costs in both human and economic aspects, and are associated with an increased risk of high blood pressure, depression, anger, anxiety, and irritability. For this reason, companies are more and more engaging in monitoring and preventing the occurrence of a stressful working environment, by addressing office vitality. This provides the further advantage of lowering the health care costs of employees while secondarily reducing absenteeism rates.

There exists already many studies in this area, which have dealt with the topic of occupational health. A common intervention in this regard is the implementation of sit-stand working stations or dynamic workstations with pedaling or walking tasks, mainly aiming to reduce the occurrence of musculoskeletal discomfort symptoms. However, a systematic review by Shrestha et al. showed that such sit-stand desks could not imply a considerable effect on working performance, and only an inconsistent effect on musculoskeletal symptoms. Moreover, walking breaks did not affect workplace sitting time whereas computer prompts to stand up had an inconsistent effect.

This indicates, that most current studies focus on promoting occupational health through physical interventions, with the main outcome being workplace sitting time and a strong focus on musculoskeletal outcomes. However, largely neglected so far are identified links of physical activity and sedentary behavior with cognition and mental health. It seems justified to assume that increasing physical activity or reducing sedentary behavior in office workers will also effect on mental health and cognition. As a way of example, the effect of a technology-based, combined physical and cognitive training, which has already been studied in various clinical settings, has only been rarely established in the context of healthy office workers. Research that analyses how this combination affects employees' health and well-being is therefore justified.

An emerging field that targets both physical and cognitive functions, are so-called exergames Exergames are games, which require the user to move his/her body to engage with a playful environment. The simultaneous cognitive task is thereby embedded in the game design, which helps to target multiple physical and cognitive functions in a combined manner. Due to the experienced enjoyment whilst playing the games, several studies reported such exergames to increase intrinsic motivation and thus adherence. Furthermore, most of the studies have shown exergames to be feasible, safe and proved them to have a high usability, as well as acceptance in geriatric, neurological, and cardiac patients. An exergame device that was developed based on this concept of combined cognitive-motor training and specifically designed for the needs of the mentioned target groups is the Dividat Senso. The ETH spin-off Dividat AG has developed this technology-based training system, with the main target of providing an optimal system for rehabilitation purposes and usage by older adults. With its hardware consisting of a pressure-sensitive step plate, surrounded by a handrail, it allows the user to interact with the software, presented on the screen in front, by the execution of steps or shifting of the body weight.

Findings from several studies in this area of cognitive-motor training have shown above all that the addition of such a cognitive training to the conventional balance and strength exercises of elderly people provide an additional positive effect on gait initiation, divided attention, and dual-task costs while walking. Due to this evidence base, the Dividat Senso was up till now mainly deployed in the field of (geriatric) research, training centers, rehabilitation clinics, and hospitals. However, with its simple operation, as well as the short intervals of the different games (2-5 minutes), the Dividat Senso could be an optimal addition to the field of occupational health, by playfully motivating employees to exercise during short work break intervals. This is supported by the study of Glazer et al. which showed that accruing physical activity in bouts of <10 minutes may already lead to a favorable influence on the general cardiometabolic risk.

The aim of this trial is, therefore, to explore whether such a combined cognitive-motor training with the Dividat Senso could be a usable and acceptable option to promote beneficial active breaks for healthy office workers. Moreover, this trial aims to assess whether this exergame training could be a way to not only interrupt the sedentary office periods with short movement bouts but also provide an optimal cognitive stimulus, leading to positive effects regarding stress and frustration levels.

ELIGIBILITY:
Inclusion Criteria:

* Provide a signed informed consent
* Aged between 18 and 65 years
* Present at min. 2 workdays a week

Exclusion Criteria:

* Severe sensory impairments (mainly visual, auditory, color blindness)
* Planned absence from work for >2 week
* Acute or unstable chronic diseases (e.g. cardiac infarction during the last year, uncontrolled high blood pressure or cardiovascular disease, uncontrolled diabetes)
* Rapidly progressing or terminal illnesses
* Chronic respiratory disease
* Condition or therapy that weakens the immune system
* Cancer
* Serious obesity > 40kg/m2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
System Usability | 6 weeks
  Score at the System Usability Scale (SUS) (for all single items and the in total) after receiving the Exergame Training for 6 weeks Higher scores imply better system usability
Technology Acceptance | 6 weeks
  Score at the Tailored Technology Acceptance Model (TAM) (for all single items and the in total) items after receiving the Exergame Training for 6 weeks Higher scores imply higher acceptance
Usability | 6 weeks
  Score at the Tailored usability questionnaire items after receiving the Exergame Training for 6 weeks
Situational Motivation Scale (SIMS) | 6 weeks
  The SIMS is a 16-item questionnaire that measures the aspects of intrinsic motivation, identified regulation, external regulation and amotivation. This brief and versatile self-report measure asks participants to rate their agree- or disagreement to predefined statements on a 7-point Likert scale.
Adherence Rate | 6 weeks
  Duration of attended exergame training sessions in relation to the duration of the recommended (2 x 10min x 6 weeks=120 minutes) sessions (in %).
Attrition | 6 weeks
  Number of participants that dropped out of the study during the exergame training intervention period.
Recruitment Rate | 6 weeks
  Number of participating employees in relation to the total number of employees working at the company and fulfilling the inclusion/exclusion criteria at the time the study took place.

SECONDARY OUTCOMES:
Changes in Mental Flexibility after 6 weeks of Exergame Training (from T1 to T2 (for G1) and from T2 to T3 (for G2) | 6 weeks of Exergame Training
  The Flexibility Test measures figural cognitive flexibility (the ability to switch between different concepts). Participants need to react as fast as possible to the presented round figure, then to the angular figure, then to the round figure and so on. Reaction times (in ms) were calculated.
Changes in Selective Attention after 6 weeks of Exergame Training (from T1 to T2 (for G1) and from T2 to T3 (for G2) | 6 weeks of Exergame Training
  The Arrow Test is used to measure selective attention and inhibition. A small grey dot in the middle of the screen needs to be fixated. On the right and left side of this grey dot, arrows appear, that point either to the right or left, in a randomized order. Steps then need to be performed as fast as possible in the direction where the arrowheads are pointing (and not the side where they are appearing). Reaction times (in ms) were calculated.
Changes in Inhibition after 6 weeks of Exergame Training (from T1 to T2 (for G1) and from T2 to T3 (for G2) | 6 weeks of Exergame Training
  The Stroop Test measures inhibition in a combination of four subtests. Four colored circles are always presented on the screen ( front=yellow, left= red, back=green, right= blue).
  During subtest (1), a square is presented in the middle, whereafter the circle with the matching color needs to be selected as fast as possible. During subtest (2), a word is presented in the middle, whereafter, the circle with the matching color needs to be selected as fast as possible. During subtest (3), word is presented in the middle, whereafter the circle needs to be selected, whose color matches the color of the letters. During subtest (4), a word appears in the middle, randomly either framed or not. If the word appears framed, the circle needs to be selected that matches the described color. If the word is unframed, the circle needs to be selected in the color of the word letters. Reaction times (in ms) were calculated in all subtests.
Changes in postural sway after 6 weeks of Exergame Training (from T1 to T2 (for G1) and from T2 to T3 (for G2) | 6 weeks of Exergame Training
  Sway Test (Senso): The Sway Test is based on the widely used Romberg Test and assesses postural control. Participants will stand on the plate with their feet shoulder-width apart and their arms extended at the front, while being standing as still as possible for 30 seconds. The test will be repeated in a second condition with closed eyes, to assess the sensory contribution to the postural control as well as in a third condition on a soft mat to assess the postural control in a more challenging environment. During these three tasks, the Center of Pressure displacement (path length in mm) is measured to evaluate participants postural control.

CONTACTS AND LOCATIONS:
Overall Officials: Eling D de Bruin, Prof., Principal Investigator — eling.debruin@hest.ethz.ch
Locations (1):
- Baryon AG, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen C, Dieterich AV, Koh JJE, Akksilp K, Tong EH, Budtarad N, Muller AM, Anothaisintawee T, Tai BC, Rattanavipapong W, Isaranuwatchai W, Rouyard T, Nakamura R, Muller-Riemenschneider F, Teerawattananon Y. The physical activity at work (PAW) study protocol: a cluster randomised trial of a multicomponent short-break intervention to reduce sitting time and increase physical activity among office workers in Thailand. BMC Public Health. 2020 Sep 1;20(1):1332. doi: 10.1186/s12889-020-09427-5. PMID 32873258
- [Background] Teychenne M, Ball K, Salmon J. Sedentary behavior and depression among adults: a review. Int J Behav Med. 2010 Dec;17(4):246-54. doi: 10.1007/s12529-010-9075-z. PMID 20174982
- [Background] Gao Y, Nevala N, Cronin NJ, Finni T. Effects of environmental intervention on sedentary time, musculoskeletal comfort and work ability in office workers. Eur J Sport Sci. 2016 Sep;16(6):747-54. doi: 10.1080/17461391.2015.1106590. Epub 2015 Nov 3. PMID 26529590
- [Background] Aegerter AM, Deforth M, Johnston V, Ernst MJ, Volken T, Luomajoki H, Brunner B, Dratva J, Sjogaard G, Elfering A, Melloh M; NEXpro collaboration group. On-site multi-component intervention to improve productivity and reduce the economic and personal burden of neck pain in Swiss office-workers (NEXpro): protocol for a cluster-randomized controlled trial. BMC Musculoskelet Disord. 2020 Jun 19;21(1):391. doi: 10.1186/s12891-020-03388-x. PMID 32560714
- [Background] Buckley JP, Hedge A, Yates T, Copeland RJ, Loosemore M, Hamer M, Bradley G, Dunstan DW. The sedentary office: an expert statement on the growing case for change towards better health and productivity. Br J Sports Med. 2015 Nov;49(21):1357-62. doi: 10.1136/bjsports-2015-094618. Epub 2015 Jun 1. PMID 26034192
- [Background] Biswas A, Oh PI, Faulkner GE, Bajaj RR, Silver MA, Mitchell MS, Alter DA. Sedentary time and its association with risk for disease incidence, mortality, and hospitalization in adults: a systematic review and meta-analysis. Ann Intern Med. 2015 Jan 20;162(2):123-32. doi: 10.7326/M14-1651. PMID 25599350
- [Background] Wilmot EG, Edwardson CL, Achana FA, Davies MJ, Gorely T, Gray LJ, Khunti K, Yates T, Biddle SJ. Sedentary time in adults and the association with diabetes, cardiovascular disease and death: systematic review and meta-analysis. Diabetologia. 2012 Nov;55(11):2895-905. doi: 10.1007/s00125-012-2677-z. Epub 2012 Aug 14. PMID 22890825
- [Background] Bhammar DM, Sawyer BJ, Tucker WJ, Gaesser GA. Breaks in Sitting Time: Effects on Continuously Monitored Glucose and Blood Pressure. Med Sci Sports Exerc. 2017 Oct;49(10):2119-2130. doi: 10.1249/MSS.0000000000001315. PMID 28514264
- [Background] Dempsey PC, Sacre JW, Larsen RN, Straznicky NE, Sethi P, Cohen ND, Cerin E, Lambert GW, Owen N, Kingwell BA, Dunstan DW. Interrupting prolonged sitting with brief bouts of light walking or simple resistance activities reduces resting blood pressure and plasma noradrenaline in type 2 diabetes. J Hypertens. 2016 Dec;34(12):2376-2382. doi: 10.1097/HJH.0000000000001101. PMID 27512975
- [Background] Falck RS, Davis JC, Liu-Ambrose T. What is the association between sedentary behaviour and cognitive function? A systematic review. Br J Sports Med. 2017 May;51(10):800-811. doi: 10.1136/bjsports-2015-095551. Epub 2016 May 6. PMID 27153869
- [Background] Thosar SS, Bielko SL, Mather KJ, Johnston JD, Wallace JP. Effect of prolonged sitting and breaks in sitting time on endothelial function. Med Sci Sports Exerc. 2015 Apr;47(4):843-9. doi: 10.1249/MSS.0000000000000479. PMID 25137367
- [Background] Elo AL, Leppanen A, Jahkola A. Validity of a single-item measure of stress symptoms. Scand J Work Environ Health. 2003 Dec;29(6):444-51. doi: 10.5271/sjweh.752. PMID 14712852
- [Background] Aldana SG. Financial impact of health promotion programs: a comprehensive review of the literature. Am J Health Promot. 2001 May-Jun;15(5):296-320. doi: 10.4278/0890-1171-15.5.296. PMID 11502012
- [Background] Davis KG, Kotowski SE. Postural variability: an effective way to reduce musculoskeletal discomfort in office work. Hum Factors. 2014 Nov;56(7):1249-61. doi: 10.1177/0018720814528003. PMID 25490805
- [Background] Schellewald V, Kleinert J, Ellegast R. Effects of two types of dynamic office workstations (DOWs) used at two intensities on cognitive performance and office work in tasks with various complexity. Ergonomics. 2021 Jun;64(6):806-818. doi: 10.1080/00140139.2020.1862308. Epub 2020 Dec 23. PMID 33289621
- [Background] Shrestha N, Kukkonen-Harjula KT, Verbeek JH, Ijaz S, Hermans V, Pedisic Z. Workplace interventions for reducing sitting at work. Cochrane Database Syst Rev. 2018 Jun 20;6(6):CD010912. doi: 10.1002/14651858.CD010912.pub4. PMID 29926475
- [Background] Healy GN, Eakin EG, Lamontagne AD, Owen N, Winkler EA, Wiesner G, Gunning L, Neuhaus M, Lawler S, Fjeldsoe BS, Dunstan DW. Reducing sitting time in office workers: short-term efficacy of a multicomponent intervention. Prev Med. 2013 Jul;57(1):43-8. doi: 10.1016/j.ypmed.2013.04.004. Epub 2013 Apr 15. PMID 23597658
- [Background] Meekes W, Stanmore EK. Motivational Determinants of Exergame Participation for Older People in Assisted Living Facilities: Mixed-Methods Study. J Med Internet Res. 2017 Jul 6;19(7):e238. doi: 10.2196/jmir.6841. PMID 28684385
- [Background] Stanmore EK, Mavroeidi A, de Jong LD, Skelton DA, Sutton CJ, Benedetto V, Munford LA, Meekes W, Bell V, Todd C. The effectiveness and cost-effectiveness of strength and balance Exergames to reduce falls risk for people aged 55 years and older in UK assisted living facilities: a multi-centre, cluster randomised controlled trial. BMC Med. 2019 Feb 28;17(1):49. doi: 10.1186/s12916-019-1278-9. PMID 30813926
- [Background] Zheng L, Li G, Wang X, Yin H, Jia Y, Leng M, Li H, Chen L. Effect of exergames on physical outcomes in frail elderly: a systematic review. Aging Clin Exp Res. 2020 Nov;32(11):2187-2200. doi: 10.1007/s40520-019-01344-x. Epub 2019 Sep 13. PMID 31520334
- [Background] Ingadottir B, Jaarsma T, Klompstra L, Aidemark J, Askenas L, Bahat Y, Ben Gal O, Berglund A, Berglund E, Hochsmann C, Plotnik M, Trappenburg JC, Schmidt-Trucksass A, Stromberg A. Let the games begin: Serious games in prevention and rehabilitation to improve outcomes in patients with cardiovascular disease. Eur J Cardiovasc Nurs. 2020 Oct;19(7):558-560. doi: 10.1177/1474515120934058. Epub 2020 Jun 13. No abstract available. PMID 32538132
- [Background] Klompstra L, Jaarsma T, Stromberg A. Exergaming to increase the exercise capacity and daily physical activity in heart failure patients: a pilot study. BMC Geriatr. 2014 Nov 18;14:119. doi: 10.1186/1471-2318-14-119. PMID 25407612
- [Background] van het Reve E, de Bruin ED. Strength-balance supplemented with computerized cognitive training to improve dual task gait and divided attention in older adults: a multicenter randomized-controlled trial. BMC Geriatr. 2014 Dec 15;14:134. doi: 10.1186/1471-2318-14-134. PMID 25511081
- [Background] Schoene D, Valenzuela T, Toson B, Delbaere K, Severino C, Garcia J, Davies TA, Russell F, Smith ST, Lord SR. Interactive Cognitive-Motor Step Training Improves Cognitive Risk Factors of Falling in Older Adults - A Randomized Controlled Trial. PLoS One. 2015 Dec 16;10(12):e0145161. doi: 10.1371/journal.pone.0145161. eCollection 2015. PMID 26673919
- [Background] Fang Q, Ghanouni P, Anderson SE, Touchett H, Shirley R, Fang F, Fang C. Effects of Exergaming on Balance of Healthy Older Adults: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Games Health J. 2020 Feb;9(1):11-23. doi: 10.1089/g4h.2019.0016. Epub 2019 Dec 3. PMID 31800322
- [Background] Glazer NL, Lyass A, Esliger DW, Blease SJ, Freedson PS, Massaro JM, Murabito JM, Vasan RS. Sustained and shorter bouts of physical activity are related to cardiovascular health. Med Sci Sports Exerc. 2013 Jan;45(1):109-15. doi: 10.1249/MSS.0b013e31826beae5. PMID 22895372
- [Background] Borsci S, Federici S, Lauriola M. On the dimensionality of the System Usability Scale: a test of alternative measurement models. Cogn Process. 2009 Aug;10(3):193-7. doi: 10.1007/s10339-009-0268-9. Epub 2009 Jun 30. PMID 19565283
- [Background] Rebsamen S, Knols RH, Pfister PB, de Bruin ED. Exergame-Driven High-Intensity Interval Training in Untrained Community Dwelling Older Adults: A Formative One Group Quasi- Experimental Feasibility Trial. Front Physiol. 2019 Aug 7;10:1019. doi: 10.3389/fphys.2019.01019. eCollection 2019. PMID 31440168
- [Background] Konstantinidis EI, Billis AS, Mouzakidis CA, Zilidou VI, Antoniou PE, Bamidis PD. Design, Implementation, and Wide Pilot Deployment of FitForAll: An Easy to use Exergaming Platform Improving Physical Fitness and Life Quality of Senior Citizens. IEEE J Biomed Health Inform. 2016 Jan;20(1):189-200. doi: 10.1109/JBHI.2014.2378814. PMID 26731797
- [Background] Potthoff T, de Bruin ED, Rosser S, Humphreys BK, Wirth B. A systematic review on quantifiable physical risk factors for non-specific adolescent low back pain. J Pediatr Rehabil Med. 2018;11(2):79-94. doi: 10.3233/PRM-170526. PMID 30010152
- [Background] Knols RH, Fischer N, Kohlbrenner D, Manettas A, de Bruin ED. Replicability of Physical Exercise Interventions in Lung Transplant Recipients; A Systematic Review. Front Physiol. 2018 Jul 20;9:946. doi: 10.3389/fphys.2018.00946. eCollection 2018. PMID 30079028
- [Background] Li J, Theng YL, Cheong WL, Hoo YF, Ngo MD. Exergames for the corporate wellness program in Singapore: An investigation of employees' acceptance via watching Kinect video. Digit Health. 2016 Jun 17;2:2055207616654578. doi: 10.1177/2055207616654578. eCollection 2016 Jan-Dec. PMID 29942559
- [Background] van Tulder M, Furlan A, Bombardier C, Bouter L; Editorial Board of the Cochrane Collaboration Back Review Group. Updated method guidelines for systematic reviews in the cochrane collaboration back review group. Spine (Phila Pa 1976). 2003 Jun 15;28(12):1290-9. doi: 10.1097/01.BRS.0000065484.95996.AF. PMID 12811274
- [Background] Shikiar R, Halpern MT, Rentz AM, Khan ZM. Development of the Health and Work Questionnaire (HWQ): an instrument for assessing workplace productivity in relation to worker health. Work. 2004;22(3):219-29. PMID 15156087
- [Background] Moore CG, Carter RE, Nietert PJ, Stewart PW. Recommendations for planning pilot studies in clinical and translational research. Clin Transl Sci. 2011 Oct;4(5):332-7. doi: 10.1111/j.1752-8062.2011.00347.x. PMID 22029804